CLINICAL TRIAL: NCT06940778
Title: LIQUID BIOPSY FOCUSING ON CIRCULATING TUMOR CELLS (CTC) AND CIRCULATING TUMOR DNA (CTDNA) AS A PRECISION MEDICINE TOOL IN GASTROINTESTINAL TUMORS
Brief Title: LIQUID BIOPSY FOCUSING ON CIRCULATING TUMOR CELLS AND CIRCULATING TUMOR DNA AS PRECISION MEDICINE IN GASTROINTESTINAL TUMORS
Acronym: BLENTI
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital do Coracao (Other)
Collaborators: Fundação Amaral Carvalho, Brazil (Unknown)
Responsible Party: Sponsor
Other Study IDs: BLENTI; 84562324.0.1001.0060 (Registry Identifier: CONEP); CONEP (Registry Identifier: Conselho Nacional de Saúde)
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cancer of Rectum; Cancer of Pancreas; Cancer of Stomach
Keywords: locally advanced rectal cancer; locally advanced and metastatic pancreas cancer; locally advanced and metastatic gastric cancer; circulating tumor cells; circulating tumor DNA; liquid biopsy
MeSH Terms: conditions — Rectal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood will be collected and circulating tumor cells and circulating tumor DNA will be isolated and analysed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Interventions — no interventions

SUMMARY:
This is a prospective, observational, multicenter cohort study. Our main objective is to to evaluate the use of CTCs and ctDNA with prognostic factors in locally advanced rectal tumors treated with total neoadjuvant therapy (TNT), recently adopted as clinical practice, and to analyze the functionality of CTCs and ctDNA in the follow-up of locally advanced and metastatic pancreatic and gastric tumors.

Secondary objectives:

* To verify the influence of CTC and ctDNA kinetics on the response to treatment of the three tumors;
* To correlate RAD23B/TYMS findings and CTC kinetics with DFS in locally advanced rectal tumors;
* To correlate HER-2 and PDL-1 expression in CTCs in gastric cancer with progression-free and overall survival;
* To verify the correlation between EGFR methylation in ctDNA of metastatic gastric tumors and PFS and OS;
* Correlate KRAS mutations in ctDNA in locally advanced pancreatic and rectal cancer with progression-free and overall survival;
* Compare the mutational profile of the primary tumor with that of the main components of the liquid biopsy (CTCs and ctDNA), in the three disease scenarios.

DETAILED DESCRIPTION:
To evaluate CTCs we will isolate cells from blood of patients by ISET method (Rarecells, France). The DNA from CTCs will be evaluated by digital PCR (Qiagen). Also, the ctDNA. Patients will be evaluated three times ( before the beginning of therapy, 6 and 12 months later. The study will be only observational. Patients will be followed by clinical and images exams.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

• Age ≥ 18 years;

For locally advanced rectal cancer:

* Patients with histological confirmation of adenocarcinoma of the distal rectum who are candidates for sphincter preservation and undergoing TNT, a long-course CRT regimen, followed by CT (5-FU + consolidation oxaliplatin);
* Tumors with a location that requires rectal amputation, except for very early tumors (cT1N0);
* Absence of distant metastases (M0).

For locally advanced or metastatic stomach cancer:

* Patients with histological confirmation of adenocarcinoma of the stomach or esophagogastric junction (EGJ) (cT2-4, cN0-3, M0-1) who have not undergone any previous treatment for the disease, surgical or systemic;
* Patients who will undergo the following treatments:

  1. (T2 to T4, N+ and M0): 4 cycles of FLOT, surgery, + 4 cycles of FLOT (5-Fluorouracil, Oxaliplatin and Docetaxel);
  2. Initial cases: T2 to T4 N0: Surgery followed by adjuvant chemotherapy: CAPOX (capecitabine + oxaliplatin) or FOLFOX (5-Fluorouracil + capecitabine) - 8 cycles;
  3. Initially unresectable T4N3: If PDL1+ and CPS > 5: CT (FOLFOX or XELOX) + nivolumab. If HER-2 + XELOX or FOLOFX + transtuzumab - after 8 cycles evaluate resectability;
  4. Metastatic disease: if HER2 negative - XELOX or FOLFOX with Nivolumab or pembrolizumab. If HER2 positive XELOX or FOLFOX with trastuzumab + pembrolizumab.

For localized or metastatic pancreatic cancer:

* Patients with histologically confirmed pancreatic adenocarcinoma (cT1-4, N0-2, M0-1) who have not undergone any prior surgical or systemic treatment for the disease.
* Patients who will undergo the following treatments:

  1. T1 to T3, N0 to N2 - resectable: Surgery followed by 12 cycles of FOLFIRINOX (oxaliplatin, 5-fluorouracil and irinotecan)
  2. Borderline resectable: Neoadjuvant chemotherapy with FOLFIRINOX for 8 cycles and surgery
  3. Unresectable disease - locally advanced: FOLFIRINOX for 12 cycles or Gemcitabine + nanoparticle paclitaxel for 8 cycles

Exclusion Criteria:

* Mid-rectum tumors or tumors with microsatellite instability.
* Stomach tumors or early EGJ (cT1N0)
* Patients who have undergone prior treatment or any surgical intervention in the last 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: brazilian population
Sampling Method: Probability Sample
Enrollment: 273 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
disease free survival | from baseline (day 1) until the date of first documented progression , assessed up to 24months
  from the diagnosis of advanced disease to disease progression

SECONDARY OUTCOMES:
overall survival | from the day one until the date of death from any cause, assessed up to 30 months
  from the diagnosis of advanced or metastatic disease to death

CONTACTS AND LOCATIONS:
Overall Officials: Ludmilla T.D. Chinen, PhD, Principal Investigator — Hospital do Coracao; LUDMILLA T.D. CHINEN, PhD, Principal Investigator — Hcor Biobank Coordinator
Locations (1):
- Hcor, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
we can share protocols and redecap data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: start date: jan-2025 end date: dec 2026
Access Criteria: researchers
URL: https://servicos3.hcor.com.br/redcap

REFERENCES:
- [Background] Abdallah EA, Braun AC, Flores BCTCP, Senda L, Urvanegia AC, Calsavara V, Fonseca de Jesus VH, Almeida MFA, Begnami MD, Coimbra FJF, da Costa WL Jr, Nunes DN, Dias-Neto E, Chinen LTD. The Potential Clinical Implications of Circulating Tumor Cells and Circulating Tumor Microemboli in Gastric Cancer. Oncologist. 2019 Sep;24(9):e854-e863. doi: 10.1634/theoncologist.2018-0741. Epub 2019 Mar 7. PMID 30846515
- [Background] Silva VSE, Abdallah EA, Flores BCT, Braun AC, Costa DJF, Ruano APC, Gasparini VA, Silva MLG, Mendes GG, Claro LCL, Calsavara VF, Aguiar Junior S, de Mello CAL, Chinen LTD. Molecular and Dynamic Evaluation of Proteins Related to Resistance to Neoadjuvant Treatment with Chemoradiotherapy in Circulating Tumor Cells of Patients with Locally Advanced Rectal Cancer. Cells. 2021 Jun 18;10(6):1539. doi: 10.3390/cells10061539. PMID 34207124
- [Background] Tarazona JGR, Abdallah EA, Flores BCT, Braun AC, Camillo CMC, Marchi FA, Ruano APC, Chinen LTD. MIR-203A-3P AND MMP-2 PROTEINS ARE HIGHLY EXPRESSED IN CIRCULATING TUMOR CELLS FROM PATIENTS WITH PANCREATIC CARCINOMA. Arq Bras Cir Dig. 2022 Jan 31;34(4):e1628. doi: 10.1590/0102-672020210002e1628. eCollection 2022. PMID 35107490
- See also: we work with liquid biopsy since 2011, with many papers published in solid and mesenchymal tumors. — https://orcid.org/orcid-search/search?searchQuery=0000-0001-7890-842
- Available data/document: Study Protocol: blenti — https://hcor.com.br — blenti